CLINICAL TRIAL: NCT06431503
Title: Effect of Tok-Sen Massage for Non-specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUH112-REC1-132
Record Dates: First submitted 2024-05-22; First posted 2024-05-28 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Non-specific Chronic Low Back Pain
Keywords: Tok-Sne massage; pressure massage; low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tok-Sen massage (Experimental): Tok-Sen massage uses a mallet to hit a wooden wedge to produce impact and sound.
  Interventions: Other: Tok-Sen Massage
- Pressure massage (Active Comparator): Pressure massage uses the wooden wedge to press.
  Interventions: Other: Pressure Massage

INTERVENTIONS:
Other: Tok-Sen Massage — Press the wedge and tapping: the strength for pressing the wedge is 1000g±50g, the height for mallet free fall(instead of beating by arm)10cm±2cm. For Pressure massage, the strength for pressing the wedge is 1500g±50g.
  Arms: Tok-Sen massage
Other: Pressure Massage — Press the wedge: the strength for pressing the wedge is 1500g±50g,
  Arms: Pressure massage

SUMMARY:
The purpose of this clinical trial was to find out whether Tok Sen massage (a massage method with wooden instruments from northern Thailand) is more effective than pressure massage in relieving pain and improving quality of life in participants with chronic low back pain. The main questions it aims to answer are:

Can Tok Sen Massage Relieve Chronic Lower Back Pain? Can Tok Sen massage improve the quality of life of patients with chronic low back pain? Researchers compared Tok Sen massage with pressure massage, which works on low back pain, to see if it could treat chronic low back pain.

Participants will:

Receive Tok Sen massage or pressure massage every week for 1 month. Questionnaires and flexion measurements before and after each massage. After the massage session, fill out the online questionnaire once a month for three months.

DETAILED DESCRIPTION:
Low back pain is the world's leading cause of global productivity loss and the leading cause of years lost with disability (YLDs), with a high prevalence of 28%-42% among those aged 40 to 69 years. The prevalence of different occupations in Taiwan ranges from 35% to 90%; according to the summary of the National Health Insurance Database results report: "The annual prevalence of low back pain is 14% to 45%, and 70% to 85% of people in their lifetime Suffering from low back pain. "Most people who experience low back pain cannot identify the specific source of the injury, and up to 90% of low back pain is non-specific. Approximately 85% of patients with low back pain cannot obtain accurate pathological anatomy diagnosis. Tok-Sen Massage is a kind of folk therapy in northern Thailand, specializing in musculoskeletal system diseases. This trial selected Pressure Massage as an active control for evaluating the effectiveness of two massage methods in improving low back pain.

This is an open-label and randomized controlled trial. Patients aged 20-69 years old with non-specific chronic low back pain were randomized divided into two different groups. 7 people in the Tok-Sen Massage group received a 40-minute intervention once a week for a total of 4 times, and 7 people the Pressure Massage group received a 40-minute intervention once a week for a total of 4 times.

Massage area are on the bladder meridian on the back and the spleen, liver and kidney meridian of the lower limbs.

The evaluation methods are: 1. Oswestry Disability Index (ODI) (baseline and after three interventions), 2. Visual Analogue Scale (VAS)before and after each massage, 3. Trunk flexibility test. before and after each massage.

ELIGIBILITY:
Inclusion Criteria:

* chronic low back pain for more than 3 months
* diagnosis of non-specific low back pain

Exclusion Criteria: -

* Spinal surgery history
* Joint disease
* Pregnancy
* Cancer
* Systemic disease
* Mental disease
* Bone Mass Measurement less than

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-11-11 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Pain relieving from Visual analogue scale | From enrollment to the end of 4 times treatments at 4 weeks
  Pain was assessed using the "Pain Visual Analogue Scale" (P-VAS), which is a self-assessment scale consisting of a 10 cm horizontal line anchored on both sides. The endpoint on the left represents "no pain." , the endpoint on the right represents "severe pain". Subjects can mark their pain level on this line based on how they feel. The distance from the position of the subject's mark to the left is the measurement result. The data range is from 0 mm to 100 mm.
  The degree of pain reduction(1%-100%, more percentage is more effective)
The Oswestry Disability Index | From enrollment to the end of follow up at 3 months
  Disability assessment uses the Oswestry Disability Index (ODI). The development of ODI was initiated by John O'Brien in 1976.
  These 10 items are respectively the degree of pain and the impact of pain on self-care, lifting heavy objects, walking ability, sitting ability, standing ability, sleep, social life, sex life and travel. Each option has 6 alternatives. The answer is scored from 0 to 5, with 0 being no pain at all and not affecting life, and 5 being extreme pain causing severe disability, so the "ODI score" ranges from 0 to 50. The calculation method of "ODI disability value": "Euclidean disability index" = (actual score/total number of questions answered × 5) × 100%. For example, all answers to 10 questions are: (actual score/50) × 100%; answer Question 9 is (actual score/45) × 100% (57, 62).

SECONDARY OUTCOMES:
Forward bend fingertip-to-floor distance | From enrollment to the end of 4 times treatments at 4 weeks
  Fingertip to Floor: The subject puts his feet and knees together, and while standing, slowly bends forward as much as possible, trying to touch the floor. The tester does not need to immobilize the pelvis, so the test allows for movement of the hip joint. Use a tape measure to measure the vertical distance from the subject's middle finger to the floor at the end of the movement.
Left and right side bending fingertip-to-floor distance subtraction | From enrollment to the end of 4 times treatments at 4 weeks
  Lateral Fingertip to Floor: The subject is in an upright position, with his back flat against the wall, his feet shoulder-width apart, and his hands hanging freely by his side. Ask the subject to bend his body to the side as much as possible , and keep back and shoulders flat against the wall, knees on both sides straight, and feet flat on the ground. When reach the end of the side bend, mark the distance of finger tip to floor.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chen Lee, M.D. & Ph.D., Study Director — China Medical University, China
Locations (1):
- China Medical University Hospital, Taichung, North Dist, Taiwan

REFERENCES:
- [Background] Snook SH. Self-care guidelines for the management of nonspecific low back pain. J Occup Rehabil. 2004 Dec;14(4):243-53. doi: 10.1023/b:joor.0000047427.21710.07. PMID 15638255
- [Background] Farooque M. Specific and nonspecific low back pain-mind the gap and its impact in clinical practice: opinion of a recovering interventional spine physiatrist. Spine J. 2023 Aug;23(8):1101-1107. doi: 10.1016/j.spinee.2023.04.011. Epub 2023 Apr 27. No abstract available. PMID 37116719
- [Background] Knezevic NN, Candido KD, Vlaeyen JWS, Van Zundert J, Cohen SP. Low back pain. Lancet. 2021 Jul 3;398(10294):78-92. doi: 10.1016/S0140-6736(21)00733-9. Epub 2021 Jun 8. PMID 34115979
- [Background] Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2940-52; discussion 2952. doi: 10.1097/00007632-200011150-00017. PMID 11074683
- [Background] Maher C, Underwood M, Buchbinder R. Non-specific low back pain. Lancet. 2017 Feb 18;389(10070):736-747. doi: 10.1016/S0140-6736(16)30970-9. Epub 2016 Oct 11. PMID 27745712
- [Background] Balague F, Mannion AF, Pellise F, Cedraschi C. Non-specific low back pain. Lancet. 2012 Feb 4;379(9814):482-91. doi: 10.1016/S0140-6736(11)60610-7. Epub 2011 Oct 6. PMID 21982256
- [Background] Chenot JF, Greitemann B, Kladny B, Petzke F, Pfingsten M, Schorr SG. Non-Specific Low Back Pain. Dtsch Arztebl Int. 2017 Dec 25;114(51-52):883-890. doi: 10.3238/arztebl.2017.0883. PMID 29321099
- [Background] Qaseem A, Wilt TJ, McLean RM, Forciea MA; Clinical Guidelines Committee of the American College of Physicians; Denberg TD, Barry MJ, Boyd C, Chow RD, Fitterman N, Harris RP, Humphrey LL, Vijan S. Noninvasive Treatments for Acute, Subacute, and Chronic Low Back Pain: A Clinical Practice Guideline From the American College of Physicians. Ann Intern Med. 2017 Apr 4;166(7):514-530. doi: 10.7326/M16-2367. Epub 2017 Feb 14. PMID 28192789
- [Background] GBD 2017 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 354 diseases and injuries for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1789-1858. doi: 10.1016/S0140-6736(18)32279-7. Epub 2018 Nov 8. PMID 30496104
- [Background] Merritt JL, McLean TJ, Erickson RP, Offord KP. Measurement of trunk flexibility in normal subjects: reproducibility of three clinical methods. Mayo Clin Proc. 1986 Mar;61(3):192-7. doi: 10.1016/s0025-6196(12)61848-5. PMID 3945120
- [Background] Chen S, Chen M, Wu X, Lin S, Tao C, Cao H, Shao Z, Xiao G. Global, regional and national burden of low back pain 1990-2019: A systematic analysis of the Global Burden of Disease study 2019. J Orthop Translat. 2021 Sep 10;32:49-58. doi: 10.1016/j.jot.2021.07.005. eCollection 2022 Jan. PMID 34934626
- [Background] Raja SN, Carr DB, Cohen M, Finnerup NB, Flor H, Gibson S, Keefe FJ, Mogil JS, Ringkamp M, Sluka KA, Song XJ, Stevens B, Sullivan MD, Tutelman PR, Ushida T, Vader K. The revised International Association for the Study of Pain definition of pain: concepts, challenges, and compromises. Pain. 2020 Sep 1;161(9):1976-1982. doi: 10.1097/j.pain.0000000000001939. PMID 32694387
- [Background] Shafshak TS, Elnemr R. The Visual Analogue Scale Versus Numerical Rating Scale in Measuring Pain Severity and Predicting Disability in Low Back Pain. J Clin Rheumatol. 2021 Oct 1;27(7):282-285. doi: 10.1097/RHU.0000000000001320. PMID 31985722
- [Background] Klineberg E, Mazanec D, Orr D, Demicco R, Bell G, McLain R. Masquerade: medical causes of back pain. Cleve Clin J Med. 2007 Dec;74(12):905-13. doi: 10.3949/ccjm.74.12.905. PMID 18183841
- [Background] Meucci RD, Fassa AG, Faria NM. Prevalence of chronic low back pain: systematic review. Rev Saude Publica. 2015;49:1. doi: 10.1590/S0034-8910.2015049005874. Epub 2015 Oct 20. PMID 26487293
- [Background] Foster NE, Anema JR, Cherkin D, Chou R, Cohen SP, Gross DP, Ferreira PH, Fritz JM, Koes BW, Peul W, Turner JA, Maher CG; Lancet Low Back Pain Series Working Group. Prevention and treatment of low back pain: evidence, challenges, and promising directions. Lancet. 2018 Jun 9;391(10137):2368-2383. doi: 10.1016/S0140-6736(18)30489-6. Epub 2018 Mar 21. PMID 29573872
- [Result] Langevin HM, Sherman KJ. Pathophysiological model for chronic low back pain integrating connective tissue and nervous system mechanisms. Med Hypotheses. 2007;68(1):74-80. doi: 10.1016/j.mehy.2006.06.033. Epub 2006 Aug 21. PMID 16919887
- [Result] Hartvigsen J, Hancock MJ, Kongsted A, Louw Q, Ferreira ML, Genevay S, Hoy D, Karppinen J, Pransky G, Sieper J, Smeets RJ, Underwood M; Lancet Low Back Pain Series Working Group. What low back pain is and why we need to pay attention. Lancet. 2018 Jun 9;391(10137):2356-2367. doi: 10.1016/S0140-6736(18)30480-X. Epub 2018 Mar 21. PMID 29573870
- [Result] Traeger AC, Buchbinder R, Elshaug AG, Croft PR, Maher CG. Care for low back pain: can health systems deliver? Bull World Health Organ. 2019 Jun 1;97(6):423-433. doi: 10.2471/BLT.18.226050. Epub 2019 Apr 30. PMID 31210680